CLINICAL TRIAL: NCT02560246
Title: Maternal Gut Microbiome (MGM) Study of Diet, the Gut Microbiome and Preterm Birth
Acronym: MGM
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: March of Dimes (Other)
Responsible Party: Sponsor
Other Study IDs: 822218
Record Dates: First submitted 2015-09-23; First posted 2015-09-25 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Preterm Birth
Keywords: Microbiome
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Collect stool, maternal blood, cord blood, and placenta from women with preterm and term labor in order to investigate whether diet and gut microbiome play a role in preterm birth.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Preterm Labor: Singleton pregnancy between 20 0/7 36 6/7 weeks gestational age who is admitted with PTL or cervical insufficiency (Equal or greater than 2 cm dilated) or PPROM
- Term Labor: Admitted to the hospital with spontaneous labor (regular contractions, cervical dilation) or spontaneous rupture of membranes

SUMMARY:
The purpose of this study is to determine whether diet and the gut microbiome play a role in spontaneous preterm birth (SPTB), namely delivery of the fetus prior to 37 weeks gestation.

DETAILED DESCRIPTION:
While dietary guidelines about intake of specific nutrients in pregnant women are well-established, surprisingly little is known about dietary eating patterns or nutritional risk factors for SPTB.

In data from two large nationally-representative European studies, SPTB was predicted by a western diet, a finding confirmed by a smaller cohort in Australia. In a small cohort in Poland, intake of short- and medium-chain fatty acids was lower in women who had SPTB, and the placental-fetal transport of fatty acids was significantly different in SPTB cases. Furthermore, more than a single serving daily of either artificially-sweetened or sugar-sweetened beverages was also linked to SPTB. Low blood biomarker levels of antioxidant nutrients (ascorbic, vitamin E)7 and nutrients with an established anti-inflammatory role in health (omega 3 fatty acids,8 vitamin D9-11) have been suggested as potential nutrient modulators of SPTB. While these are very interesting findings, they do not explain whether these food patterns prevail in an urban U.S. population or why SPTB occurs. Furthermore, none of these potentially modifiable diet associations has been examined in the context of the entire series of physiological systems operating during pregnancy, namely diet, the gut microbiome, maternal plasma metabolome, placenta, and cord blood.

There is biological rationale to assume that dietary components could modify the gut microbiome and the maternal plasma metabolome during pregnancy. Artificial sweeteners induce glucose intolerance through an alternation in the gut microbiota. Chronic ingestion of sugar-sweetened beverages also results in similar plasma metabolic abnormalities (gut microbiome measures were not reported). In animal models of high fat diet feeding (similar to western diet), addition of N3FA ameliorated the gut dysbiosis and reduced endotoxin production. Furthermore, in healthy volunteers, the investigators have recently linked typical dietary intake patterns with the gut microbiome. Dietary patterns of high protein and animal fat intake were predominantly associated with Bacteroides enterotypes, while carbohydrate intake was associated with Prevotella. While the microbiome composition changes rapidly after change in diet, the enterotype identity is resilient over time. The investigators followed these findings with another study comparing the extreme diets of vegans (no animal products) to the more typical mixed western diet pattern of omnivores, and extended the analytical approaches to include assessment of the plasma metabolome. By observing the microbiome and metabolome, the investigators were clearly able to distinguish with 91% accuracy whether a subject was vegan or omnivore. Furthermore, the investigators could determine metabolomic characteristics that were contributed by gut bacterial metabolism, but only in subjects with high plant food intake. These findings in healthy volunteers raise the possibility that gut microbial populations could interact with maternal tissues or plasma to produce an inflammatory state that might result in preterm parturition. Indeed, the alteration of the gut microbiota observed in the third trimester of pregnancy and its effects on host metabolism are supportive of this notion.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women receiving care in University of Pennsylvania Health System
* Between 16-24 weeks gestation

Exclusion Criteria:

* Multiple gestation
* Fetal chromosomal abnormality or major fetal anomaly
* Intrauterine fetal demise
* Maternal HIV
* Chronic kidney disease
* Transplant
* Prior weight loss surgery
* Vegan diet
* Chronic use of immunosuppresive medications or steriods

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women will be recruited from three locations: Penn ObGyn Associates, Helen O. Dickens Clinic, and Maternal Fetal Medicine at 2000 Courtyard. Potential subjects will be identified from clinical schedules and will be pre-screened in EPIC for eligibility. They may be approached during a clinical visit, or the research team may call them prior to or after a scheduled visit to introduce the study. Women can be enrolled anytime between the confirmation of pregnancy and 24 weeks/0 days gestation. For convenience, research visits can be conducted at the time of a scheduled clinical visit, or at a separate time.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-05-04 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2017-08-29 (Actual)

PRIMARY OUTCOMES:
Preterm Birth | At time of delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States